CLINICAL TRIAL: NCT03202381
Title: A Pilot Phase IV Study to Evaluate Variation in Bone Mineral Density, Lean and Fat Body Mass Index Measured by Dual-energy X-ray Absorptiometry in Patients With Prostate Cancer Without Bone Metastasis Treated With Degarelix
Brief Title: Phase IV Study to Evaluate Bone Mineral Density in No-bone Metastatic Prostate Cancer Treated With Degarelix
Acronym: BLADE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Alessandro Antonelli, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NP2540-BLADE
Record Dates: First submitted 2017-06-12; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: Androgen deprivation therapy; GnRH antagonist
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Degarelix (Experimental)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Degarelix (Firmagon®) will be administered as a subcutaneous injection in the abdominal region every 28 days, in according to the following schedule:
  * Starting dose: 240 mg administered as two consecutive subcutaneous injections of 120 mg each (2 x 3 mL injections).
  * Maintenance dose: 80 mg administered as one subcutaneous injection of 80 mg (1 x 4 mL injection).
  Treatment will be continued till clinically indicated or till disease progression.

SUMMARY:
The aim of this phase IV interventional study is to evaluate variation in bone mineral density and lean and fat body composition in patients with prostate cancer without bone metastasis, treated with Degarelix. These variations are evaluated at time 0 (before starting androgen deprivation therapy with Degarelix) and after 12 months of therapy by dual-energy X-ray absorptiometry (DXA scan).

DETAILED DESCRIPTION:
Gonadotropin-releasing hormone (GnRH) agonists decrease bone mineral density (BMD) and increase fracture risk in men with prostate carcinoma. GnRH agonists also increase fat mass and decrease lean body mass. These treatment-related changes in body composition may contribute to fatigue, emotional distress, and decreased quality of life. Whereas the consequences of initial GnRH agonist on BMD and body composition are well characterized, less is known regarding the effects of GnRH antagonists. At the best of our knowledge the changes in body composition induced by Degarelix in prostate cancer patients has never been explored. Dual-energy X-ray absorptiometry (DXA) is a reliable and accurate method to determine the changes in body composition in patients with prostate cancer (PCa) undergoing androgen deprivation therapy (ADT).

The change in body composition is a major determinant of increased morbidity and mortality induced by ADT and DXA provides the most precise measure of body composition. This study is designed to obtain explorative information on changes in bone mineral density, fat body mass and lean body mass by DXA scan after administration of Degarelix. These preliminary data compared with historical data of patients submitted to GnRH agonists could provide a rationale for a subsequent prospective randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* male outpatients, aged 18 or older, willing and able to provide written informed consent;
* histological diagnosis of prostate carcinoma;
* more than 6-month survival prospect;
* no bone metastases as assessed by bone scintigraphy;
* eligibility to ADT with Degarelix in the opinion of the clinical investigator.

Exclusion Criteria:

* patients with absolute or relative contraindication for prescription of Degarelix. In particular:
* hypersensitivity towards any component of Firmagon®
* patients who receive concomitant medications that might prolong the QT interval, in particular class I A (such as quinidine, procainamide, disopyramide,) or class III antiarrhythmics (such as amiodarone, sotalol, dofetilide, ibutilide)
* patients with history of or risk factors for Torsades de Pointes
* patients who take either methadone or moxifloxacin or antipsychotic
* patients with alteration in electrolyte blood levels (such as sodium, potassium, calcium and magnesium)
* patients with severe kidney and/or liver dysfunctions;
* concomitant bone metabolic disease, such as Paget's disease, primary hyperparathyroidism or chronic hypercortisolism, as recorded by medical history;
* renal failure (baseline serum creatinine more than 1.5 mg/dl);
* prior hormonal treatment;
* prior or concomitant treatment with bisphosphonates or other drugs known to affect bone metabolism (for example steroids, calcitonin);
* patients participating in an interventional clinical trial in which any treatment or follow-up is mandated;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Changes in fat body mass | 12 months
  To determine changes in fat body mass after 12 months Degarelix administration.

SECONDARY OUTCOMES:
changes in bone mineral density | 12 months
  to assess changes in bone mineral density after 12 months of therapy;
changes in lean body mass | 12 months
  to assess changes in lean body mass after 12 months of therapy;
changes in fasting serum lipids | 12 months
  to assess changes in fasting serum lipids after 12 months of therapy;
changes in bone turn-over markers | 12 months
  to assess changes in bone turn-over markers after 12 months of therapy;
changes in insulin sensitivity | 12 months
  to assess changes in insulin sensitivity after 12 months of therapy;
changes in serum follicle stimulating hormone (FSH) levels | 12 months
  to assess changes in serum FSH levels after 12 months of therapy;

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Department of Urology, university Hospital Spedali Civili di Brescia, Brescia, Italy

REFERENCES:
- [Background] Smith MR. Changes in fat and lean body mass during androgen-deprivation therapy for prostate cancer. Urology. 2004 Apr;63(4):742-5. doi: 10.1016/j.urology.2003.10.063. PMID 15072892
- [Background] Eri LM, Urdal P, Bechensteen AG. Effects of the luteinizing hormone-releasing hormone agonist leuprolide on lipoproteins, fibrinogen and plasminogen activator inhibitor in patients with benign prostatic hyperplasia. J Urol. 1995 Jul;154(1):100-4. PMID 7539852
- [Background] Smith MR, Finkelstein JS, McGovern FJ, Zietman AL, Fallon MA, Schoenfeld DA, Kantoff PW. Changes in body composition during androgen deprivation therapy for prostate cancer. J Clin Endocrinol Metab. 2002 Feb;87(2):599-603. doi: 10.1210/jcem.87.2.8299. PMID 11836291
- [Background] Smith MR. Osteoporosis and other adverse body composition changes during androgen deprivation therapy for prostate cancer. Cancer Metastasis Rev. 2002;21(2):159-66. doi: 10.1023/a:1020840311573. PMID 12465755
- [Background] Smith MR, Lee H, Nathan DM. Insulin sensitivity during combined androgen blockade for prostate cancer. J Clin Endocrinol Metab. 2006 Apr;91(4):1305-8. doi: 10.1210/jc.2005-2507. Epub 2006 Jan 24. PMID 16434464
- [Background] Berruti A, Dogliotti L, Terrone C, Cerutti S, Isaia G, Tarabuzzi R, Reimondo G, Mari M, Ardissone P, De Luca S, Fasolis G, Fontana D, Rossetti SR, Angeli A; Gruppo Onco Urologico Piemontese (G.O.U.P.), Rete Oncologica Piemontese. Changes in bone mineral density, lean body mass and fat content as measured by dual energy x-ray absorptiometry in patients with prostate cancer without apparent bone metastases given androgen deprivation therapy. J Urol. 2002 Jun;167(6):2361-7; discussion 2367. PMID 11992038
- [Background] Buttigliero C, Vana F, Bertaglia V, Vignani F, Fiori C, Osella G, Porpiglia F, Tucci M, Scagliotti GV, Berruti A. The fat body mass increase after adjuvant androgen deprivation therapy is predictive of prostate cancer outcome. Endocrine. 2015 Sep;50(1):223-30. doi: 10.1007/s12020-015-0525-x. Epub 2015 Jan 15. PMID 25588772
- [Derived] Bergamini M, Dalla Volta A, Palumbo C, Zamboni S, Triggiani L, Zamparini M, Lagana M, Rinaudo L, Di Meo N, Caramella I, Bresciani R, Valcamonico F, Borghetti P, Guerini A, Farina D, Antonelli A, Simeone C, Mazziotti G, Berruti A. Relationship between circulating FSH levels and body composition and bone health in patients with prostate cancer who undergo androgen deprivation therapy: The BLADE study. Elife. 2024 Apr 24;13:e92655. doi: 10.7554/eLife.92655. PMID 38656229
- [Derived] Palumbo C, Dalla Volta A, Zamboni S, Mazziotti G, Zamparini M, Triggiani L, Borghetti P, Maffezzoni F, Bresciani R, Rinaudo L, Valcamonico F, Farina D, Magrini SM, Antonelli A, Simeone C, Berruti A. Effect of Degarelix Administration on Bone Health in Prostate Cancer Patients Without Bone Metastases. The Blade Study. J Clin Endocrinol Metab. 2022 Nov 25;107(12):3398-3407. doi: 10.1210/clinem/dgac489. PMID 35971857